CLINICAL TRIAL: NCT04069156
Title: Antiplatelet Removal and HemocompatIbility EventS With the HeartMate 3 Pump IDE Study
Brief Title: The ARIES HeartMate 3 Pump IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ABT-CIP-10305
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
Keywords: heart failure; ventricular assist device; LVAD; aspirin
MeSH Terms: conditions — Heart Failure | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized 1:1, active arm versus placebo arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, site, patient, CEC, and core lab are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): LVAD Patients on the placebo arm will be given placebo medication
  Interventions: Device: LVAD Implant; Drug: Placebo oral tablet
- Active Arm (Active Comparator): LVAD Patients on the active arm will be given 100mg Aspirin
  Interventions: Device: LVAD Implant; Drug: Aspirin 100mg

INTERVENTIONS:
Device: LVAD Implant — Subjects will undergo Heartmate 3 LVAD implant prior to randomization
Drug: Aspirin 100mg — Subjects will be randomized to either Placebo or Aspirin post implant.
  Arms: Active Arm
Drug: Placebo oral tablet — Subjects will be randomized to either Placebo or Aspirin post implant
  Arms: Placebo Arm

SUMMARY:
Prospective, randomized, double-blinded, placebo-controlled clinical investigation of advanced heart failure patients treated with the HM3 with two different antithrombotic regimens: vitamin K antagonist with aspirin versus vitamin K antagonist with placebo

DETAILED DESCRIPTION:
This clinical investigation is a prospective, randomized, double-blinded, placebo-controlled study of advanced heart failure patients treated with the HM3 with two different antithrombotic regimens: vitamin K antagonist with aspirin versus vitamin K antagonist with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will receive the HeartMate 3 per standard of care (SOC) in accordance with the approved indications for use in the country of implant.
2. Subject will receive the HeartMate 3 as their first durable VAD.
3. Subject must provide written informed consent prior to any clinical investigation related procedure.
4. In female patients of child bearing capability, subject will not be currently pregnant or breastfeeding and on appropriate contraception.

Exclusion Criteria:

1. Post-implant additional temporary or permanent mechanical circulatory support (MCS).
2. Investigator mandated antiplatelet therapy for other conditions (including mandated presence or absence of antiplatelet agent).
3. Patients who are nil per os (NPO) post-implant through day 7.
4. Subjects with a known allergy to acetylsalicylic acid (aspirin).
5. Participation in any other clinical investigation(s) involving an MCS device, or interventional investigation(s) likely to confound study results or affect study outcome.
6. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (41):
  - Baptist Health Medical Center, Little Rock, Arkansas
  - University of California, San Diego, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center - Van Ness Campus, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Miami Transplant Institute - Jackson Memorial, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Montefiore Medical Center - Moses Division, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Hospital, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Aurora Medical Group, Milwaukee, Wisconsin
- Australia (2):
  - St. Vincent's Hospital, Sydney, Darlinghurst, New
  - The Alfred Hospital, Melbourne, Victoria
- AKH - Wien, Vienna, Austria
- University of Alberta Hospital, Edmonton, Canada
- IKEM Prague, Prague, Central Bohemia, Czechia
- France (2):
  - Hopital Haut Leveque, Pessac
  - CHU Rangueil Toulouse, Toulouse
- Ospedale San Raffaele, Milan, Italy
- National Research Center for Cardiac Surgery, Astana, Kazakhstan
- Queen Elizabeth Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To be determined

REFERENCES:
- [Background] Mehra MR, Netuka I, Uriel N, Katz JN, Pagani FD, Jorde UP, Gustafsson F, Connors JM, Ivak P, Cowger J, Ransom J, Bansal A, Takeda K, Agarwal R, Byku M, Givertz MM, Bitar A, Hall S, Zimpfer D, Vega JD, Kanwar MK, Saeed O, Goldstein DJ, Cogswell R, Sheikh FH, Danter M, Pya Y, Phancao A, Henderson J, Crandall DL, Sundareswaran K, Soltesz E, Estep JD; ARIES-HM3 Investigators. Aspirin and Hemocompatibility Events With a Left Ventricular Assist Device in Advanced Heart Failure: The ARIES-HM3 Randomized Clinical Trial. JAMA. 2023 Dec 12;330(22):2171-2181. doi: 10.1001/jama.2023.23204. PMID 37950897
- [Background] Gustafsson F, Uriel N, Netuka I, Katz JN, Pagani FD, Connors JM, Jorde UP, Zimpfer D, Pya Y, Conway J, Anyanwu A, Scandroglio AM, Sulemanjee N, Atluri P, Keebler M, Selzman CH, Alexis JD, Hayward C, Henderson J, Dirckx N, Gazzola C, Mehra MR; ARIES Investigators. Aspirin and Hemocompatibility After LVAD Implantation in Patients With Atherosclerotic Vascular Disease: A Secondary Analysis From the ARIES-HM3 Randomized Clinical Trial. JAMA Cardiol. 2025 Mar 1;10(3):235-242. doi: 10.1001/jamacardio.2024.4849. PMID 39774588
- [Background] Mehra MR, Crandall DL, Gustafsson F, Jorde UP, Katz JN, Netuka I, Uriel N, Connors JM, Sood P, Heatley G, Pagani FD. Aspirin and left ventricular assist devices: rationale and design for the international randomized, placebo-controlled, non-inferiority ARIES HM3 trial. Eur J Heart Fail. 2021 Jul;23(7):1226-1237. doi: 10.1002/ejhf.2275. Epub 2021 Jul 1. PMID 34142415
- [Derived] Katz JN, Connors JM, Pagani FD, Jorde UP, Gustafsson F, Uriel N, Netuka I, Byku M, Anyanwu A, Keebler M, Nathan S, Selzman CH, Alexis JD, Sulemanjee N, Atluri P, D'Allesandro D, Porter S, Lee FS, Mehra MR; ARIES Investigators. Hemocompatibility Outcomes With Pharmacological Therapy Following LVAD Implantation: Insights From the ARIES-HM3 Trial. JACC Heart Fail. 2025 Nov 19:102769. doi: 10.1016/j.jchf.2025.102769. Online ahead of print. PMID 41258850
- [Derived] Pagani FD, Netuka I, Jorde UP, Katz JN, Gustafsson F, Connors JM, Uriel N, Soltesz EG, Ivak P, Bansal A, Bitar A, Vega JD, Goldstein D, Danter M, Pya Y, Ravichandran A, Conway J, Adler ED, Chung ES, Grinstein J, Dirckx N, Iravani B, Mehra MR. Concomitant Surgical Procedures and Aspirin Avoidance With Left Ventricular Assist Device Therapy. JACC Heart Fail. 2025 Jul;13(7):102411. doi: 10.1016/j.jchf.2025.01.017. Epub 2025 Apr 9. PMID 40208135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled and randomized 628 subjects at 51 sites. Enrollment took place between July 2020 and September 2022, with the last subject follow up concluding in August 2023.
Pre-assignment Details: The intent to treat (ITT) population consisted of all subjects randomized including follow up beyond transition to open label (n=314 in each arm).
Groups:
- Placebo Arm: Patients randomized to the placebo arm were given placebo medication.
- Aspirin Arm: Patients randomized to the aspirin arm were given aspirin medication (100mg/day).
Period: Modified Intent-to-Treat (mITT)
Arm/Group | Placebo Arm | Aspirin Arm
Started | 314 (18 patients experienced surgical events and outcomes required cessation of treatment within 14 days.) | 314 (21 patients experienced surgical events and outcomes required cessation of treatment within 14 days.)
Completed | 296 | 293
Not Completed | 18 | 21
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Transitioned to open label | 8 | 12
Period: Principal Analysis
Arm/Group | Placebo Arm | Aspirin Arm
Started | 296 | 293
Completed | 271 | 273
Not Completed | 25 | 20
Not completed — Withdrawn without primary end point event | 25 | 20

BASELINE CHARACTERISTICS:
Population: The Modified Intention to Treat Population (mITT) included all randomized subjects with the following exception:
  1. Subjects who experienced a surgical adverse event, defined as ≤14 days post-implant, requiring investigator mandated antiplatelet therapy;
  2. Subjects who expired, are transplanted, or withdrawn within 14 days of implant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Aspirin Arm | Total
Number analyzed (Participants) | 296 | 293 | 589
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.8) | 56.5 (14.4) | 57.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 61 | 133
  Male | 224 | 232 | 456
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 9 | 22
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 93 | 84 | 177
  White | 179 | 181 | 360
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 6 | 13 | 19
Heart Failure Etiology [Count of Participants; unit: Participants]
  Ischemic Cardiomyopathy | 106 | 101 | 207
  Idiopathic Cardiomyopathy | 68 | 63 | 131
  Dilated Cardiomyopathy | 86 | 81 | 167
  Other | 36 | 48 | 84
Intended Use [Count of Participants; unit: Participants]
  Bridge to Transplantation | 56 | 58 | 114
  Bridge to Candidacy for Transplantation | 46 | 50 | 96
  Destination Therapy | 180 | 174 | 354
  Bridge to Recovery | 14 | 11 | 25
INTERMACS Profile [Count of Participants; unit: Participants] — INTERMACS profiles describe the clinical profile of advanced heart failure patients who may be candidates for mechanical circulatory support. There are 7 profiles ranging from Profile 1 (most sick) to Profile 7 (least sick). Profile 1 indicates critical cardiogenic shock. Profile 2 indicates progressive decline. Profile 3 indicates stable but inotrope dependent. Profile 4 indicates resting symptoms. Profile 5 indicates exertion intolerant. Profile 6 indicates exertion limited. Profile 7 indicates advanced NYHA Class 3 (clinically stable with a reasonable level of comfortable activity).
  Participants
    1 | 12 | 18 | 30
    2 | 76 | 75 | 151
    3 | 133 | 133 | 266
    4 | 66 | 54 | 120
    5 | 6 | 8 | 14
    6 | 3 | 5 | 8
    7 | 0 | 0 | 0
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — The NYHA functional classification consists of four categories, with Class IV being the worse class.
  * Class I: No symptoms or limitation in ordinary physical activity
  * Class II: Mild symptoms and slight limitation during ordinary activity
  * Class IIIA or B: NYHA class IIIA patients experience no dyspnea at rest, while NYHA class IIIB patients experience recent dyspnea at rest. Both patient classes have marked limitations in physical activity, even with less than ordinary activity.
  * Class IV: Severe limitations, experiences symptoms even while at rest
  Participants
    Class II | 3 | 2 | 5
    Class IIIA | 27 | 29 | 56
    Class IIIB | 40 | 38 | 78
    Class IV | 226 | 224 | 450
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 251 | 248 | 499
  Other | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Powered Primary Endpoint of Survival Free of Non-surgical Major Hemocompatibility Related Adverse Events
Description: The primary end point was a composite of survival free of non-surgical major hemocompatibility related adverse events (specifically stroke, pump thrombosis, major non-surgical bleeding, and arterial peripheral thromboembolism) at 1-year post implant.
Time Frame: 12 Months
Population: The primary end point was analyzed in the principal analysis population, which excluded patients with events occurring within 14 days after LVAD implantation to avoid counting surgical complications not attributed to the treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Arm (Principal Analysis Population): Patients randomized to the placebo arm were given placebo medication.
- Aspirin Arm (Principal Analysis Population): Patients randomized to the aspirin arm were given aspirin medication (100mg/day).
Arm/Group | Placebo Arm (Principal Analysis Population) | Aspirin Arm (Principal Analysis Population)
Number analyzed (Participants) | 271 | 273
Participants | 201 | 186
Statistical Analysis 1: Comparison: Placebo Arm (Principal Analysis Population) vs Aspirin Arm (Principal Analysis Population); Test type: Non-Inferiority — The primary end point assessing non-inferiority of placebo was considered met if the lower boundary of the one-sided 97.5% confidence limit of the difference in the composite success rate between treatment arms (placebo minus aspirin) was greater than the non-inferiority margin (-10%) by the Farrington-Manning test at 12-months in the principal analysis population; p < 0.0001, Farrington-Manning risk difference; Risk Difference (RD) = 6, 97.5% CI 1-sided [lower limit -1.6]

2. Secondary Outcome: Rates of Non-surgical Major Hemorrhagic Events
Description: The rate of non-surgical hemorrhagic events were compared between the two arms of the study. Non-surgical Major Hemorrhagic events: Hemorrhagic event rate per patient year was calculated by dividing all non-surgical bleeding events and hemorrhagic stroke events by the cumulative years of study exposure.
Time Frame: Through Study Completion with a Median Follow up of 14 Months
Population: Modified Intention to Treat Population (mITT)
Measure: Number; unit: Event Per 100 Patient-Year
Groups:
- Placebo Arm (Modified Intent-to-treat Population): Patients randomized to the placebo arm were given placebo medication.
- Aspirin Arm (Modified Intent-to-treat Population): Patients randomized to the aspirin arm were given aspirin medication (100mg/day).
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Event Per 100 Patient-Year
  All Non-surgical Major Hemorrhagic events | 26.2 | 40.7
  Bleeding | 25.93 | 39.53
  Hemorrhagic Stroke | 0.27 | 0.85
  Ischemic Stroke with Hemorrhagic Conversion | 0.00 | 0.28

3. Secondary Outcome: Rates of Bleeding Events
Description: The bleeding rate was calculated by dividing the number of bleeding events by the cumulative duration of study exposure (years of support).
Time Frame: Through Study Completion with a Median Follow up of 14 Months
Population: Modified Intention to Treat Population (mITT)
Measure: Number; unit: Event Per 100 Patient-Year
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Event Per 100 Patient-Year
  All Bleeding Events | 25.92 | 39.53
  Moderate Bleeding | 8.46 | 13.65
  Severe Bleeding | 17.47 | 25.88
  GI Bleeding | 13.10 | 21.61
  Fatal Bleeding | 0.55 | 0.85

4. Secondary Outcome: Rates of Non-surgical Major Thrombotic Events
Description: The rates of non-surgical major thrombotic events was compared between the two arms of the study. The thrombotic event rate per patient year was calculated by dividing the number of non-surgical ischemic strokes, pump thrombosis and arterial peripheral thromboembolic events by the cumulative years of study exposure
Time Frame: Through Study Completion with a Median Follow up of 14 Months
Population: Modified Intention to Treat Population (mITT)
Measure: Number; unit: Event Per 100 Patient-Year
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Event Per 100 Patient-Year
  All Major Thrombotic events | 1.64 | 2.84
  Ischemic Stroke without Hemorrhagic Conversion | 1.64 | 2.56
  Device Thrombosis | 0.00 | 0.00
  Arterial Peripheral Thromboembolism | 0.00 | 0.00

5. Secondary Outcome: Rates of Stroke
Description: The stroke rate was calculated based on the number of strokes experienced by subjects, 14 days or more after device implant, and while on their treatment assignment, divided by the cumulative duration of study exposure (years of support).
Time Frame: Through Study Completion with a Median Follow up of 14 Months
Population: Modified Intention to Treat Population (mITT)
Measure: Number; unit: Event Per 100 Patient-Year
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Event Per 100 Patient-Year
  All Stroke | 1.91 | 3.70
  Debilitating Stroke (MRS>3) | 0.82 | 0.57
  Non-Debilitating Stroke (MRS<=3) | 1.09 | 3.13

6. Secondary Outcome: Survival Rates
Description: The overall survival rate was analyzed using a Kaplan-Meier analysis and the treatment groups were compared using log-rank test. Survival was calculated starting at 14 days post implant.
Time Frame: 24 Months
Population: Modified Intention to Treat Population (mITT)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Percentage of Participants | 93 | 89.7

7. Secondary Outcome: Risk of Non-Surgical Bleeding Events
Description: Risk of non-surgical bleeding events was analyzed using a Kaplan-Meier analysis. The treatment groups were compared using a log-rank test.
Time Frame: 24 Months
Population: Modified Intention to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Percentage of Participants | 30.0 | 42.4

8. Other Pre Specified Outcome: Rate of Rehospitalization
Description: This study assessed changes in the rehospitalization as a result of removal of antiplatelet therapy from the antithrombotic regimen.
Time Frame: Through Study Completion with a Median Follow up of 14 Months
Population: Modified Intention to Treat Population
Measure: Number; unit: Event Per 100 Patient-Year
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 296 | 293
Event Per 100 Patient-Year
  Hemocompatibility Related | 0.15 | 0.28
  Major Infection | 0.34 | 0.36
  Hypertension | 0.03 | 0.02
  Cardiovascular Related | 0.33 | 0.33
  Non-cardiovascular organ dysfunction | 0.06 | 0.05
  Neurologic dysfunction (excluding stroke, TIA) | 0.01 | 0.02
  Other | 0.41 | 0.42

9. Other Pre Specified Outcome: Economic Cost Implications - Total Estimated Cost for Bleeding Events (CMS Cost Basis)
Description: Cost of bleeding episodes was calculated based on a previously published economic model, adjusted for inflation using the US Bureau of Labor Statistics Medical Consumer Price Index. To ensure uniformity in care practices and relevance of the previously published model, only US subjects were included.
Time Frame: 12 Months
Population: Only US subjects were included in this analysis
Measure: Number; unit: USD
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 247 | 244
USD | 546,947 | 927,040

10. Other Pre Specified Outcome: Economic Cost Implications - Average Cost Per Bleeding Event
Description: These values were derived by dividing the total estimated cost for bleeding events by the number of events to determine the average cost per bleeding event. Consequently, a measure of dispersion is not available for these outcomes.
Time Frame: 12 Months
Population: Only US subjects were included in this analysis
Measure: Number; unit: USD
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 247 | 244
USD | 13,674 | 13,836

11. Other Pre Specified Outcome: Economic Cost Implications - Average Cost Per Study Patient Over the First-year Post-implant
Description: These values were derived by dividing the total estimated cost for bleeding events by the number of patients to obtain the average cost per study patient. Consequently, a measure of dispersion is not available for these outcomes.
Time Frame: 12 Months
Population: Only US subjects were included in this analysis
Measure: Number; unit: USD
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 247 | 244
USD | 2,214 | 3,799

12. Other Pre Specified Outcome: Economic Cost Implications - Cost of Bleeding Hospitalization for 1000 LVAD Implants Over the First-year Post-implant
Description: as for outcome 9
Time Frame: 12 Months
Population: Only US subjects were included in this analysis
Measure: Number; unit: USD/1000 implants/1 year
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
Number analyzed (Participants) | 247 | 244
USD/1000 implants/1 year | 2,214,362 | 3,799,344

ADVERSE EVENTS:
Time Frame: All adverse events occurring through study completion (median follow up of 14 months) were collected.
Description: An adverse event (AE) is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Placebo Arm (Modified Intent-to-treat Population) | Aspirin Arm (Modified Intent-to-treat Population)
All-Cause Mortality (participants affected / at risk) | 21/296 | 22/293
Serious Adverse Events (participants affected / at risk) | 208/296 | 223/293
Other Adverse Events (participants affected / at risk) | 200/296 | 181/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (Modified Intent-to-treat Population) (N=296) | Aspirin Arm (Modified Intent-to-treat Population) (N=293)
Bleeding (Blood and lymphatic system disorders) | 68 (92) | 100 (138) — Site reported event terms were used for protocol defined adverse events.
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Site reported event terms were used for protocol defined adverse events.
Cardiac Arrhythmia (Cardiac disorders) | 44 (59) | 41 (73) — Site reported event terms were used for protocol defined adverse events.
Right Heart Failure (Cardiac disorders) | 12 (14) | 6 (8) — Site reported event terms were used for protocol defined adverse events.
Hepatic Dysfunction (Hepatobiliary disorders) | 6 (6) | 4 (4) — Site reported event terms were used for protocol defined adverse events.
Major Infection (Infections and infestations) | 99 (201) | 116 (197) — Site reported event terms were used for protocol defined adverse events.
Neurologic Dysfunction (Nervous system disorders) | 25 (25) | 21 (29) — Site reported event terms were used for protocol defined adverse events.
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 14 (19) — Site reported event terms were used for protocol defined adverse events.
Renal Dysfunction (Renal and urinary disorders) | 15 (18) | 2 (3) — Site reported event terms were used for protocol defined adverse events.
Venous Thromboembolism (Vascular disorders) | 2 (2) | 3 (3) — Site reported event terms were used for protocol defined adverse events.
Hypertension (Vascular disorders) | 9 (12) | 7 (7) — Site reported event terms were used for protocol defined adverse events.
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 3 (3) | 4 (7) — Other events reported by MedDRA system organ classification.
Cardiac Disorders (Cardiac disorders) | 33 (64) | 35 (51) — Other events reported by MedDRA system organ classification.
Ear And Labyrinth Disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Other events reported by MedDRA system organ classification.
Endocrine Disorders (Endocrine disorders) | 3 (3) | 2 (2) — Other events reported by MedDRA system organ classification.
Eye Disorders (Eye disorders) | 1 (1) | 1 (1) — Other events reported by MedDRA system organ classification.
Gastrointestinal Disorders (Gastrointestinal disorders) | 24 (26) | 13 (17) — Other events reported by MedDRA system organ classification.
General Disorders And Administration Site Conditions (Gastrointestinal disorders) | 31 (39) | 24 (34) — Other events reported by MedDRA system organ classification.
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0) — Other events reported by MedDRA system organ classification.
Immune System Disorders (Immune system disorders) | 0 (0) | 1 (1) — Other events reported by MedDRA system organ classification.
Infections And Infestations (Infections and infestations) | 2 (2) | 3 (3) — Other events reported by MedDRA system organ classification.
Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 15 (16) | 17 (20) — Other events reported by MedDRA system organ classification.
Investigations (Investigations) | 14 (18) | 17 (20) — Other events reported by MedDRA system organ classification.
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 32 (40) | 33 (44) — Other events reported by MedDRA system organ classification.
Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (6) — Other events reported by MedDRA system organ classification.
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) — Other events reported by MedDRA system organ classification.
Nervous System Disorders (Nervous system disorders) | 22 (26) | 26 (34) — Other events reported by MedDRA system organ classification.
Pregnancy, Puerperium And Perinatal Conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Other events reported by MedDRA system organ classification.
Psychiatric Disorders (Psychiatric disorders) | 5 (6) | 2 (2) — Other events reported by MedDRA system organ classification.
Renal And Urinary Disorders (Renal and urinary disorders) | 11 (13) | 8 (10) — Other events reported by MedDRA system organ classification.
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 25 (35) | 24 (31) — Other events reported by MedDRA system organ classification.
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Other events reported by MedDRA system organ classification.
Social Circumstances (Social circumstances) | 0 (0) | 1 (1) — Other events reported by MedDRA system organ classification.
Surgical And Medical Procedures (Surgical and medical procedures) | 1 (1) | 1 (1) — Other events reported by MedDRA system organ classification.
Vascular Disorders (Vascular disorders) | 22 (31) | 20 (24) — Other events reported by MedDRA system organ classification.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (Modified Intent-to-treat Population) (N=296) | Aspirin Arm (Modified Intent-to-treat Population) (N=293)
Major Infection (Infections and infestations) | 94 (129) | 92 (118) — Site reported event terms were used for protocol defined adverse events.
Cardiac Arrhythmia (Cardiac disorders) | 8 (9) | 11 (12) — Site reported event terms were used for protocol defined adverse events.
Hepatic Dysfunction (Hepatobiliary disorders) | 5 (5) | 6 (6) — Site reported event terms were used for protocol defined adverse events.
Venous Thromboembolism (Vascular disorders) | 4 (4) | 4 (4) — Site reported event terms were used for protocol defined adverse events.
Bleeding (Blood and lymphatic system disorders) | 3 (4) | 1 (1) — Site reported event terms were used for protocol defined adverse events.
Renal Dysfunction (Renal and urinary disorders) | 3 (3) | 0 (0) — Site reported event terms were used for protocol defined adverse events.
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 14 (15) | 10 (11) — Other events reported by MedDRA system organ classification.
Cardiac Disorders (Cardiac disorders) | 42 (52) | 23 (33) — Other events reported by MedDRA system organ classification.
Eye Disorders (Eye disorders) | 14 (14) | 2 (2) — Other events reported by MedDRA system organ classification.
Gastrointestinal Disorders (Gastrointestinal disorders) | 21 (27) | 18 (22) — Other events reported by MedDRA system organ classification.
General Disorders And Administration Site Conditions (General disorders) | 34 (43) | 21 (26) — Other events reported by MedDRA system organ classification.
Hepatobiliary Disorders (Hepatobiliary disorders) | 6 (7) | 1 (1) — Other events reported by MedDRA system organ classification.
Infections And Infestations (Infections and infestations) | 5 (5) | 3 (3) — Other events reported by MedDRA system organ classification.
Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 20 (25) | 24 (31) — Other events reported by MedDRA system organ classification.
Investigations (Investigations) | 25 (51) | 29 (54) — Other events reported by MedDRA system organ classification.
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 43 (61) | 33 (36) — Other events reported by MedDRA system organ classification.
Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 19 (21) | 15 (15) — Other events reported by MedDRA system organ classification.
Nervous System Disorders (Nervous system disorders) | 40 (45) | 26 (29) — Other events reported by MedDRA system organ classification.
Psychiatric Disorders (Psychiatric disorders) | 16 (21) | 9 (11) — Other events reported by MedDRA system organ classification.
Renal And Urinary Disorders (Renal and urinary disorders) | 19 (29) | 8 (12) — Other events reported by MedDRA system organ classification.
Reproductive System And Breast Disorders (Reproductive system and breast disorders) | 5 (5) | 1 (1) — Other events reported by MedDRA system organ classification.
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 27 (31) — Other events reported by MedDRA system organ classification.
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 15 (15) | 9 (9) — Other events reported by MedDRA system organ classification.
Vascular Disorders (Vascular disorders) | 36 (44) | 39 (49) — Other events reported by MedDRA system organ classification.

LIMITATIONS AND CAVEATS:
We excluded patients with early surgical complications or those that required mechanical support devices in addition to the implanted LVAD, or when investigators deemed aspirin therapy necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT04069156/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT04069156/SAP_001.pdf